CLINICAL TRIAL: NCT02688218
Title: Testing and Tuning a Multiparameter Exercise Detection Algorithm
Brief Title: Exercise Detection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joseph El Youssef, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 15452
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Type 1 Diabetes
Keywords: exercise; artificial pancreas; hypoglycemia; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic First, Resistance Second (Experimental): Subjects will complete three 15 minute periods of aerobic exercise, with 10 minute recovery between each period. This will be followed by 5-15 minute periods of up to 7 activities of daily living with an additional 20 minute period of resistance exercise, such as straight leg raises.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Resistance Exercise
- Resistance First, Aerobic Second (Experimental): Subjects will complete 5-15 minute periods of up to 7 activities of daily living with an additional 20 minute period of resistance exercise, such as straight leg raises. This will be followed by three 15 minute periods of aerobic exercise, with 10 minute recovery between each period.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Exercise for three 15 minute periods, with 10 minute rests between each period, and exercise intensity will vary between periods to achieve different energy expenditures, which may be determined based on VO2 measurements.
Behavioral: Resistance Exercise — Subjects will perform 5-15 minutes of up to 7 different activities of daily living, followed by 20 minutes of resistance exercise, such as straight leg raises.

SUMMARY:
The risk of hypoglycemia in individuals with type 1 diabetes increases considerably during exercise. As a result, many patients with type 1 diabetes experience fear of and reluctance to pursue physical activity, in order to avoid the discomforting symptoms associated with hypoglycemia. The bi-hormonal artificial pancreas, a device used for automatic delivery of insulin and glucagon subcutaneously to subjects with type 1 diabetes, is paving the way to revolutionize the management of this disease. The investigator's group has recently completed a study of the bi-hormonal artificial pancreas system during exercise, suggesting reduced hypoglycemia around the exercise period. In order to prepare for a future home study, the ability to detect, grade, and classify physical activity so as to appropriately adjust system parameters is vital in helping to prevent exercise induced hypoglycemia in the home setting.

This study is designed to collect 3-axis accelerometry data and heart rate data during a variety of different home activities, as well as during formal exercise in both healthy subjects and subjects with type 1 diabetes. Additionally, the investigators will observe the change in glucose levels before and after exercise in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
The artificial pancreas, a device used for automatic delivery of insulin and glucagon subcutaneously to subjects with type 1 diabetes, is paving the way to revolutionize the management of this disease. Already, the benefit of improved glycemic control compared to current open-loop pump therapy has been demonstrated in several trials. The investigator's group has shown that artificial pancreas algorithm dual hormone system effectively manages blood glucose in a clinic setting and the investigators have specifically shown great progress using glucagon to reduce hypoglycemic episodes outside of exercise. The investigators most recent inpatient study, as yet unpublished, shows that adjusting insulin and glucagon delivery during closed loop treatment, after announcing exercise, effectively reduces mean time below a glucose level of 70 mg/dl when compared to closed loop control without adjustments. The investigators utilized initial open-loop data from this study to help devise dosing changes for the artificial pancreas algorithm.

In order to prepare for a future home study, the ability to detect, grade, and classify physical activity so as to appropriately adjust system parameters is vital in helping to prevent exercise induced hypoglycemia in the home setting. Currently, our closed-loop system transmits heart rate and accelerometry outputs from a Zephyrlife BioPatch monitoring device to a Nexus 5 smart phone master controller via Bluetooth. The algorithm then converts the heart rate and accelerometry data into modified estimated energy expenditure - accounting for age, weight, height, sex, resting and sitting heart rates - to determine if exercise is present. However, further data collection is needed to hone the specificity and sensitivity of the detection algorithm to account for a wide variety of subject characteristics and activities.

This study is designed to collect 3-axis accelerometry data and heart rate data during a variety of different home activities, as well as during formal exercise, which included aerobic exercise (on a calibrated treadmill) and resistance exercise (straight-leg raises or equivalent) in healthy subjects as well as subjects with type 1 diabetes. Optionally VO2 data from a portable VO2 mask will be obtained. The data collected will be used to further enhance our algorithm that, in future closed-loop studies, will detect exercise and automatically trigger algorithmic adjustments to reduce exercise-related hypoglycemia during and after exercise in individuals with type 1 diabetes.

ELIGIBILITY:
TYPE 1 DIABETIC SUBJECT CRITERIA

Inclusion criteria:

1. Male or female subjects 21 to 45 years of age with a diagnosis of T1D for at least 6 months on an insulin pump.
2. Physically active on a regular basis, i.e. at least 3 days of scheduled physical activity per week and willing to perform approximately 60 minutes of exercise (as determined by the investigator after reviewing the subjects activity level).
3. Willingness to follow all study procedures.
4. Willingness to sign informed consent and HIPAA documents.

Exclusion criteria:

a. Pregnancy or Lactation: i. For women of childbearing potential, there is a requirement for a negative urine pregnancy test. b. Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary. c. Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as report by the OHSU laboratory). d. Hematocrit of less than or equal to 34%. e. History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. f. Adrenal insufficiency. g. Any active infection. h. Known or suspected abuse of alcohol, narcotics, or illicit drugs (except marijuana use).

i. Seizure disorder. j. Active foot ulceration. k. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication. l. Major surgical operation within 30 days prior to screening. m. Use of an investigational drug within 30 days prior to screening. n. Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus). o. Bleeding disorder, treatment with warfarin, or platelet count below 50,000. p. Current administration of oral or parenteral corticosteroids. q. Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer). r. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen. s. Beta blockers or non-dihydropyridine calcium channel blockers. t. A positive response to any of the questions from the Physical Activity Readiness Questionnaire, see Appendix A. u. Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort. v. Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

HEALTHY SUBJECT CRITERIA

Inclusion Criteria:

1. Male or female subjects 21 to 45 years of age.
2. Physically active on a regular basis, i.e. at least 3 days of scheduled physical activity per week and willing to perform approximately 60 minutes of exercise (as determined by the investigator after reviewing the subjects activity level).
3. Willingness to follow all study procedures.
4. Willingness to sign informed consent and HIPAA documents.

Exclusion criteria:

1. Pregnancy or Lactation: For women of childbearing potential, there is a requirement for a negative urine pregnancy test.
2. Any history or evidence of renal insufficiency, adrenal insufficiency, liver disease or anemia.
3. A history of cerebrovascular disease or coronary artery disease (or angina) regardless of the time since occurrence.
4. Congestive heart failure, New York Heart Association (NYHA) any class.
5. Diagnosis of 1st, 2nd or 3rd degree heart block or any arrhythmia judged by the investigator to be exclusionary.
6. Any condition which, in the opinion of the investigator, makes it difficult to engage in vigorous physical activity.
7. Any active infection.
8. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
9. Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator).
10. Active malignancy, except basal cell or squamous cell skin cancers.
11. Major surgical operation within 30 days prior to screening.
12. Seizure disorder.
13. Bleeding disorder, or treatment with warfarin.
14. Use of any chronic medications.
15. Use of an investigational drug within 30 days prior to screening.
16. Any reason the principal investigator deems exclusionary.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph El Youssef, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castle JR, Engle JM, El Youssef J, Massoud RG, Yuen KC, Kagan R, Ward WK. Novel use of glucagon in a closed-loop system for prevention of hypoglycemia in type 1 diabetes. Diabetes Care. 2010 Jun;33(6):1282-7. doi: 10.2337/dc09-2254. Epub 2010 Mar 23. PMID 20332355
- [Background] Jacobs PG, El Youssef J, Castle J, Bakhtiani P, Branigan D, Breen M, Bauer D, Preiser N, Leonard G, Stonex T, Ward WK. Automated control of an adaptive bihormonal, dual-sensor artificial pancreas and evaluation during inpatient studies. IEEE Trans Biomed Eng. 2014 Oct;61(10):2569-81. doi: 10.1109/TBME.2014.2323248. Epub 2014 May 13. PMID 24835122
- [Background] Jacobs PG, El Youssef J, Castle JR, Engle JM, Branigan DL, Johnson P, Massoud R, Kamath A, Ward WK. Development of a fully automated closed loop artificial pancreas control system with dual pump delivery of insulin and glucagon. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:397-400. doi: 10.1109/IEMBS.2011.6090127. PMID 22254332
- [Background] Jacobs PG, Resalat N, El Youssef J, Reddy R, Branigan D, Preiser N, Condon J, Castle J. Incorporating an Exercise Detection, Grading, and Hormone Dosing Algorithm Into the Artificial Pancreas Using Accelerometry and Heart Rate. J Diabetes Sci Technol. 2015 Oct 5;9(6):1175-84. doi: 10.1177/1932296815609371. PMID 26438720
- Available data/document: Study Protocol: STUDY00015452 — http://eirb.ohsu.edu — Institutionally reviewed and accepted protocol for this study.

RESULTS

PARTICIPANT FLOW:
Period: First Exercise Intervention (2 Hours)
Arm/Group | Aerobic First, Resistance Second | Resistance First, Aerobic Second
Started | 24 | 6
Completed | 24 | 6
Not Completed | 0 | 0
Period: Washout (30 Minutes)
Arm/Group | Aerobic First, Resistance Second | Resistance First, Aerobic Second
Started | 24 | 6
Completed | 24 | 6
Not Completed | 0 | 0
Period: Second Exercise Intervention (2 Hours)
Arm/Group | Aerobic First, Resistance Second | Resistance First, Aerobic Second
Started | 24 | 6
Completed | 24 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic First, Resistance Second | Resistance First, Aerobic Second | Total
Number analyzed (Participants) | 24 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 6 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.1) | 31.4 (4.7) | 31.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 3 | 17
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 6 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 21 | 6 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Type 1 Diabetes [Count of Participants; unit: Participants] | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Sensor Glucose in Subjects With Type 1 Diabetes
Description: The mean change in sensor glucose before and after both exercise periods (aerobic and resistance) during the study visit, obtained from Dexcom G4 sensors in the subjects with type 1 diabetes.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aerobic Exercise | Resistance Exercise
Number analyzed (Participants) | 7 | 7
mg/dL | -26.4 (41.1) | 12.0 (28.5)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Aerobic Exercise: Subjects will complete three 15 minute periods of aerobic exercise, with 10 minute recovery between each period.
  Aerobic Exercise: Exercise for three 15 minute periods, with 10 minute rests between each period, and exercise intensity will vary between periods to achieve different energy expenditures, which may be determined based on VO2 measurements.
- Resistance Exercise: Subjects will complete 5-15 minute periods of up to 7 activities of daily living with an additional 20 minute period of resistance exercise, such as straight leg raises.
  Resistance Exercise: Subjects will perform 5-15 minutes of up to 7 different activities of daily living, followed by 20 minutes of resistance exercise, such as straight leg raises.
Arm/Group | Aerobic Exercise | Resistance Exercise
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT02688218/Prot_SAP_000.pdf